CLINICAL TRIAL: NCT03954574
Title: Pulmonary Hemodynamics During Exercise - Research Network
Acronym: PEX-NET
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: European Respiratory Society (Other)
Responsible Party: Sponsor
Other Study IDs: 30-437 ex 17/18
Record Dates: First submitted 2019-03-14; First posted 2019-05-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Circulation Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective patient cohort
  Interventions: Diagnostic Test: assessment of pulmonary hemodynamics during exercise by right heart catheterization
- Prospective patient cohort
  Interventions: Diagnostic Test: assessment of pulmonary hemodynamics during exercise by right heart catheterization

INTERVENTIONS:
Diagnostic Test: assessment of pulmonary hemodynamics during exercise by right heart catheterization — all patients undergo right heart catheterization during exercise due to clinical reasons. Results of this and other Routine clinical tests will be included in the registry

SUMMARY:
The purpose of this Clinical Research Collaboration is to investigate the prognostic implications of pulmonary hemodynamics during exercise based on a large scale multi-centre approach by using retrospective and prospective analysis of hemodynamic data.

ELIGIBILITY:
Inclusion Criteria:

* Patients (females and males; age: above 18yrs) with intermediate or high echocardiographic probability of PH and/or unexplained dyspnea, and/or associated conditions for PAH as clinical indication for RHC at rest and exercise
* Written informed consent of participating subjects after being fully briefed (for prospective analysis)

Exclusion Criteria:

* Patients with incomplete hemodynamic data at rest or exercise
* Patients without sufficient follow-up data (information on survival / lung transplantation)
* advanced tumour disease or other diseases with a short life expectancy, except pulmonary vascular diseases
* advanced heart failure with pulmonary arterial wedge pressure (PAWP) > 18 mmHg at rest
* uncontrolled systemic arterial hypertension (RR values > 160/100 mmHg at rest)
* FEV1<50% predicted
* TLC<60% predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (females and males; age: above 18yrs) with intermediate or high echocardiographic probability of PH and/or unexplained dyspnea, and/or associated conditions for PAH as clinical indication for right heart catheterization at rest and exercise
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who die during observation | 6 years
  The investigators aim to assess the prognostic relevance of pulmonary hemodynamics during exercise as assessed by right heart catheterization by using a multi-centre approach and to identify independent predictors of adverse events. Separate data sets will be analysed for the retrospective and prospective Evaluation.
Number of Participants undergoing lung Transplantation during observation | 6 years
  Occurrences of lung transplantations

SECONDARY OUTCOMES:
Number of Participants being hospitalized during observation | 6 years
  Number of hospitalizations
Number of Participants who develop pulmonary Hypertension as assessed by right heart catheterization | 6 years
  Diagnosis of pulmonary hypertension
Number of Participants with newly initiated pulmonary arterial Hypertension medication during observation | 6 years
  Evaluation of medication initiations

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Study Chair — Medical University of Graz; Philippe Herve, MD, Study Chair — Centre Chirugical Marie Lannelongue
Locations (32):
- United States (8):
  - University of Arizona, Banner University Medical Center, Phoenix, Arizona
  - University of California, Los Angeles, Lung & Heart-Lung Transplant and Pulmonary Hypertension Programs, David Geffen School of Medicine, Los Angeles, California
  - Johns Hopkins Hospital, Advanced HF, MCS, Transplant Cardiology, Baltimore, Maryland, USA, Baltimore, Maryland
  - Massachusetts General Hospital, Cardiology Division and Pulmonary Unit, Boston, Massachusetts
  - Harvard Medical School, Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota Medical School, Division of Cardiology, Department of Medicine, Lillehei Heart Institute Minneapolis, Minnesota, USA, Minneapolis, Minnesota
  - Mayo Clinic, Division of Cardiovascular Diseases, Department of Medicine, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina
- Royal Prince Alfred Hospital, Respiratory Medicine, Camperdown, Australia
- Medical University of Graz, Graz, Austria
- Free University of Brussels, Faculty of Medicine, Physiology, Brussels, Belgium
- University of São Paulo Medical School, São Paulo, Brazil
- Department of Cardiology, Aarhus University Hospital, Denmark, Aarhus, Denmark
- France (4):
  - Université de Lorraine, Nancy
  - Centre Chirurgical Marie Lannelongue, Thoracic and Vascular Surgery, Paris
  - Centre de Référence de l'Hypertension Pulmonaire, Université ParisSud - Université Paris-Saclay, Hôpital Bicêtre, Assistance Publique Hôpitaux de Paris, Paris
  - Sorbonne Universités, Neurophysiologie respiratoire expérimentale et clinique, Paris
- Germany (5):
  - University of Cologne, Klinik III fuer Innere Medizin, Cologne
  - Justus-Liebig-University Giessen, Department of Internal Medicine, Giessen
  - University of Greifswald, Greifswald
  - Thorax Clinic Heidelberg, Centre for Pulmonary Hypertension, Heidelberg
  - Academic Teaching Hospital of the Julius Maximilian University of Würzburg, Würzburg
- Italy (2):
  - University of Bologna, Bologna
  - University of Rome La Sapienza, Cardiovascular and Respiratory Sciences, Roma
- VU Medisch Centrum, Pulmonology, Amsterdam, Netherlands
- Otwock Medical Center of Postgraduate Education, Department of Pulmonary Circulation and Thromboembolic Diseases, Otwock, Poland
- Barcelona Hospital Clínic, Pneumologia, Barcelona, Spain
- University Hospital of Zurich, Internal Medicine, Zurich, Switzerland
- United Kingdom (4):
  - Scottish Pulmonary Vascular Unit, Glasgow
  - Imperial College, NHS Healthcare NHS Trust, National Pulmonary Hypertension Service, London
  - Royal Brompton Hospital, London
  - Royal Hallamshire Hospital, Sheffield Pulmonary Vascular Disease Unit, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided